CLINICAL TRIAL: NCT02221921
Title: Clinical Evaluation of the Safety and Performance of the MicroPort's Transcatheter Aortic Valve and Delivery System for Treatment of Severe Aortic Stenosis
Brief Title: Safety and Efficacy Study of MicroPort's Transcatheter Aortic Valve and Delivery System for TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0000SYV; MicroPort Medical (Registry Identifier: MicroPort Medical)
Record Dates: First submitted 2014-08-14; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Calcification
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve, Calcification of

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MicroPort's Transcatheter Aortic Valve and Delivery System (Experimental): single arm with intervention that percutaneous implantation of the MicroPort's Transcatheter Aortic Valve and Delivery System
  Interventions: Device: MicroPort's Transcatheter Aortic Valve and Delivery System

INTERVENTIONS:
Device: MicroPort's Transcatheter Aortic Valve and Delivery System

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the MicroPort's Valve and delivery system for transcatheter aortic valve implantation (TAVI) in severe aortic stenosis who are considered unsuitable for Surgical Valve Replacement.

DETAILED DESCRIPTION:
1. Evaluate the performance, safety and clinical benefit of MicroPort's aortic valve prosthesis and delivery system in intervention by peripheral artery.
2. The study Continuous observe 12 months of safety and efficacy. Approximately 89 patients are recruited in the study with native aortic valve stenosis which are considered unsuitable for Surgical Valve Replacement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, male or non pregnant women;
* Senile degenerative aortic valve stenosis with echocardiography derived criteria: mean gradient ≥ 40 mmHg, or jet velocity ≥ 4.0 m/s, or an aortic valve area (AVA) of < 1.0 cm2 (or AVA index < 0.6 cm2/m2)
* Symptomatic due to aortic valve stenosis as demonstrated by NYHA (New York Heart Association) Functional Class ≥ II
* Expectation of life>12 months
* Calcific aortic stenosis, which is suitable for transcatheter aortic valve implantation anatomically
* is evaluated by at least two cardiovascular physicians, and they agreed that medical factors precluding operation suitable for surgery (the probability of death or serious, irreversible morbidity exceeded 50%)
* The subject agreed to comply follow-up evaluation

Exclusion Criteria:

* Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment
* aortic valve is a congenital unicuspid valve, or is non-calcified.
* Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days
* Implanted any heart valve prosthesis, prosthetic valve ring, severe（>3＋）mitral valve insufficiency
* Blood dyscrasia such as leukopenia (WBC < 3×109/L), acute anemia (Hgb < 90 g/L), thrombocytopenia (PLT < 50×109/L), bleeding diathesis, or history of coagulopathy.
* Untreated clinically significant coronary artery disease requiring revascularization
* Hemodynamic instability requiring mechanical cardiac assist or mechanical hemodynamic support devices
* Need for emergency surgery for any reason
* Hypertrophic cardiomyopathy with or without obstruction
* Severe ventricular dysfunction with LVEF (Left ventricular ejection fraction) < 20%
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active peptic ulcer or upper gastro-intestinal bleeding within the prior 3 months
* A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, Nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated.
* Native aortic annulus size < 17 mm or> 29 mm.
* Patient refuses aortic valve replacement surgery.
* Cerebrovascular Accident (CVA) within 6 months, including TIA (transient ischemic attack).
* Renal insufficiency (creatinine > 3.0 mg/dL) and/or end stage renal disease requiring chronic dialysis.
* Life expectancy < 12 months
* Significant abdominal or thoracic aorta disease, including aneurysm, marked tortuosity (hyperacute bend), aortic arch atheroma, narrowing of the abdominal aorta (especially with calcification and surface irregularities), or severe "unfolding" and tortuosity of the thoracic aorta
* Iliofemoral vessel characteristics that would preclude safe placement of 16F to 19F introducer sheath such as severe obstructive calcification, severe tortuosity
* Active bacterial endocarditis or other active infections.
* Bulky calcified aortic valve leaflets in close proximity to coronary ostia
* severe incapacitating dementia.
* Currently participating in an investigational drug or another device study that has not reached its primary endpoint.
* Researchers identify that the patients with poor compliance who cannot be completed in accordance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
All cause mortality or major stroke at 12 months. | 12 months

SECONDARY OUTCOMES:
MACCE(major adverse cardiovascular and cerebrovascular events) | 30 days, 3, 6 and 12 months
  MACCE is defined as a composite of:
  * Myocardial infarction (MI)
  * Hemorrhage
  * renal failure
  * vascular complications
  * block
  * ventricular arrhythmias
Device success | 7 days post-operation
  Device success is defined as
  * The device successfully enter the vascular approach, transport and release
  * The valve is placed in the correct anatomical position
  * The valve achieve the expected effect (mean aortic pressure < 20mmHg or peak velocity < 3m/s, with no severe aortic regurgitation or paravalvular leakage)
Valve performance | 30 days, 3, 6 and 12 months
  Valve performance means:
  * Transvalvular mean gradient
  * Effective orifice area
  * Degree of aortic valve regurgitation (transvalvular and paravalvular)
The improvement of heart function | 30 days, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JunBo Ge, Medical Doctor, Professor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China